CLINICAL TRIAL: NCT05428358
Title: Incremental Value of Magnetic Resonance Imaging in Selection of Pancreatic Cancer Patients for Surgery (MAGIPAC): A Randomized Clinical Trial.
Brief Title: Incremental Value of Magnetic Resonance Imaging in Selection of Pancreatic Cancer Patients for Surgery
Acronym: MAGIPAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Rigshospitalet, Denmark (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MAGIPAC
Record Dates: First submitted 2022-06-16; First posted 2022-06-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer; Pancreatic Neoplasm; Liver Metastases
Keywords: magnetic resonance imaging
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative MRI (Experimental): MRI before surgery.
  Interventions: Diagnostic Test: Preoperative MRI

INTERVENTIONS:
Diagnostic Test: Preoperative MRI — Preoperative MRI performed between outpatient visit at the surgical clinic and scheduled date of resection

SUMMARY:
The aim of the study is to examine the incremental value of using magnetic resonance imaging (MRI) in addition to computed tomography (CT) in the diagnostic workup of pancreatic cancer patients.

DETAILED DESCRIPTION:
The aim of the study is to examine the incremental value of using magnetic resonance imaging (MRI) in addition to computed tomography (CT) in the diagnostic workup of pancreatic cancer patients. We will conduct a nationwide, prospective clinical trial to examine the incremental value of using MRI for identification of liver metastases in pancreatic cancer patients.

ELIGIBILITY:
Inclusion criteria:

* Pancreatic cancer patients considered to have a locally resectable or borderline resectable tumor by the local hepato-pancreato-biliary multidisciplinary team board
* No liver metastases on CT
* At least 18 years old and able to provide informed consent
* Expected pancreatic ductal adenocarcinoma based on CT scan

Exclusion criteria:

* Metastatic disease
* Prior receipt of neoadjuvant chemotherapy or downstaging/-sizing treatment
* Comorbidity rendering major surgery unfeasible (inoperable)
* No informed consent
* Unable to undergo MRI (Kidney insufficiency (eGFR < 60 ml/min/1.73 m2 body surface ar-ea); Claustrophobia; Cardiac pacemaker)
* Postoperative histology other than adenocarcinoma of pancreato-biliary origin.
* MRI with liver-specific contrast performed during standard workup.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in treatment strategy | 1 week
  Change in treatment strategy from intended curative resection to other treatment based on MRI scan

SECONDARY OUTCOMES:
Liver metastases | 1 week
  Proportion of patients who had liver metastases detected on MRI
Surgery | 1 month
  Proportion of patients who made it to surgery/exploration
Resection | 1 month
  Proportion of patients in each arm who had a pancreatic resection performed
Intraoperatively detected liver metastases | 1 month
  Proportion of patients with intraoperatively detected liver metastases not seen on either CT or MRI.
Overall survival (1-year) | 1 year
  1-year overall survival.
Overall survival (3-year) | 3 years
  3-year overall survival.
Recurrence-free survival | 3 years
  Recurrence-free survival according to final treatment strategy.
Healthcare costs | 3 years
  Healthcare costs in patients with change of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Mortensen, MD, DMSc, Study Chair — Aarhus University Hospital; Jakob Kirkegård, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No
Due to Danish law, no individual-level data can be shared.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT05428358/Prot_SAP_002.pdf